CLINICAL TRIAL: NCT05917249
Title: Efficacy of Capacitive-Resistive Noninvasive Radiofrequency in Improving Perfusion Index and Attenuating Diabetic Neuropathic Pain; A Pre-post Study
Brief Title: Efficacy of Noninvasive Radiofrequency in Attenuating Diabetic Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ms-399-2022
Record Dates: First submitted 2023-06-05; First posted 2023-06-23 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional (Experimental)
  Interventions: Device: Capacitive-Resistive Noninvasive Radiofrequency

INTERVENTIONS:
Device: Capacitive-Resistive Noninvasive Radiofrequency — The two passive plates were under the back of the patient. The active capacitive plates of the machine (CAPENGERY, C200, Spain) will be applied initially for 20 minutes over the sole of both feet, with the machine adjusted on the A-thermal mode (37 oC). During the remaining 20 minutes, active capacitive plates are relocated over femoral vessels at the femoral triangle with the machine adjusted on the frank thermal mode (41 oC).
  Other Names: TECAR

SUMMARY:
Peripheral neuropathy increases the prevalence of diabetic foot ulcers following a decrease in foot sensation. Therefore, the treatment of this disorder is very important.

DETAILED DESCRIPTION:
The current study aimed to investigate the efficacy of TECAR therapy on lower limb perfusion index (PI) and to evaluate the efficacy of TECAR therapy in improving the peripheral vascularity, reducing foot pain, and improving the tactile sensation of the soles in diabetic peripheral neuropathy (DPN) patients. twenty three diabetic neuropathy patients were included in the study and underwent 12 sessions of Capacitive TECAR therapy over one month. Pain, tactile sensation of the sole and PI were evaluated at the start and after each session till the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Type II DM with DPN (grade I-II) in lower limbs
* Duration of DM>5 years
* Visual Analog Scale (VAS) ≥3 in the feet
* Sensory impairments in the lower extremities

Exclusion Criteria:

* Patient with previous stenting or surgical intervention of lower limb arterial system.
* Patients with previous history of DVT.
* Pregnancy
* Diabetic infectious wound
* Cardiac pacemaker presence
* Severe liver and kidney dysfunction or history of heart and lung disease.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change of the perfusion index at the end of the first session compared to baseline readings. | 40 minutes
  the perfusion index readings will be taken before the first session and set as baseline reading and after the first session and the change will be calculated.The Masimo SET "Mighty-Sat Fingertip Pulse Oximetry" (Masimo Corporation, Irvine, CA, USA model 9900) was attached to the big toe of each patient. the reading will be the the mean of three measurements of perfusion index (PI) taken at one-minute intervals.

SECONDARY OUTCOMES:
Visual Analogue Scale | 2 months
  Patient defines the degree of pain on a visual scale without numeric values, while the values are visible on the back side for the registrar where 0 indicates no pain and 10 indicates the most unbearable pain. The test was performed before intervention, after each session and one month after the end of all twelve sessions.
Tactile sensation of the sole | 2 months
  Tactile sensation of the sole using Semmes-Weinstein monofilament 5.07/10 g. the test will be performed after each session.
Analgesic effect | 2 months
  * Analgesic effect after each session; will be evaluated using the four grades of WHO evaluation criteria for pain relief:
  * Complete remission (CR)
  * Partial remission (PR)
  * Mild remission (MR)
  * No response (NR).
The total remission rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelrauof, MD, Principal Investigator — Cairo University; Waleed Al-Hamimy, MD, Principal Investigator — Cairo University
Locations (1):
- Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niajalili M, Sedaghat M, Reazasoltani A, Akbarzade Baghban AR, Sadat Naimi S. [Effect of Capacitive Tecar Therapy on Foot Pain and Tactile Sensation in Patients With Type 2 Diabetes (Persian)]. Archives of Rehabilitation. 2020; 21(3):304-319. https://doi.org/10.32598/RJ.21.3.60.5
- [Background] Tashiro Y, Hasegawa S, Yokota Y, Nishiguchi S, Fukutani N, Shirooka H, Tasaka S, Matsushita T, Matsubara K, Nakayama Y, Sonoda T, Tsuboyama T, Aoyama T. Effect of Capacitive and Resistive electric transfer on haemoglobin saturation and tissue temperature. Int J Hyperthermia. 2017 Sep;33(6):696-702. doi: 10.1080/02656736.2017.1289252. Epub 2017 Feb 19. PMID 28139939